CLINICAL TRIAL: NCT04821219
Title: Establishing a Platform for Personalized Approach to the Management of Pancreatic Adenocarcinoma Using Patient-Derived Tumoroids
Brief Title: Personalized Management of Pancreatic Adenocarcinoma Using Patient-Derived Tumoroids
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study PI no longer at Institution
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Panagiotis Z. Anastasiadis, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-010804
Record Dates: First submitted 2021-02-23; First posted 2021-03-29 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Pancreas Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tumoroid generation (Experimental): Single arm, including all the patients enrolled to generate tumor models
  Interventions: Other: Treatment prediction PDT platform

INTERVENTIONS:
Other: Treatment prediction PDT platform — PDT will be generated and response to various chemotherapies and radiation will be investigated. Actionable targets will be identified and response to the target drug will be assessed and compared to the conventional treatment options.

SUMMARY:
This study is designed to prospectively investigate the feasibility of establishing patient-derived tumoroids (PDT) as a platform for a personalized approach for response prediction and guide optimal neoadjuvant and/or adjuvant approach. PDT will be investigated to determine drug sensitivity, predict the response to chemotherapy agents and radiation therapy, and validate this response in treated patients, and to establish the feasibility of PDT as a platform for a personalized approach to guide multimodality treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age.
* Have an ECOG Performance Status of ≤ 2.
* No evidence of distant metastasis on imaging.
* Histologic or cytologic proven adenocarcinoma of the pancreas.
* Providing informed consent prior to enrollment in the trial.

Exclusion Criteria:

* Failure to obtain additional core needle biopsies for generating PDTs.
* Females who are pregnant or plan to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of the successful establishment of pancreatic patient-derived tumoroids (PDT) | 2 years

SECONDARY OUTCOMES:
Drug sensitivity and response prediction of chemotherapy agents in PDT | 2 years
  the PDT response to the treatment with conventional regimens for treatment of (pancreatic adenocarcinoma (PDAC) and other approved treatments based on pharmacogenomic analysis. Treatment response will be assessed with viability assays.
Drug sensitivity and response prediction of radiation therapy in PDT | 2 years
  the PDT response to the treatment with radiation with or without radiosensitizers. Treatment response will be assessed with viability assays.
PDT validation with a comparative analysis of patients' response to neoadjuvant chemotherapy and radiation | 2 years
  Response evaluation according to imaging based on RECIST (Response Evaluation Criteria in Solid Tumors) criteria, biochemical response in CA19-9 and pathologic response in the surgical specimen vs. PTD response in the corresponding neoadjuvant regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Anastasiadis, PhD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials